CLINICAL TRIAL: NCT06940999
Title: Revolutionizing Scar Evaluation: An Innovative Image-Based Method for Extensibility Assessment
Brief Title: An Innovative Image-Based Method for Extensibility Assessment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Ahmed Elsayeh, Asst. Prof. Dr., Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P.T.REC/012/005678
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Hypertrophic Scar
Keywords: Image-based assessment; Scar extensibility assessment.
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Intervention Model Description: Mixed-method design combining quasi-experimental and instrument validation approaches
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Traditional physical therapy group (Experimental): This study uses a mixed-method design combining a quasi-experimental, single-group pre-post intervention with a methodological validation approach.
  Participants will receive a standardized physical therapy protocol targeting scar contracture. After intervention, scar extensibility will be measured using traditional tools (Vancouver Scar Scale, tonometer) and a newly developed image-based method. The image-based method will be tested for:
  * Reliability (test-retest, inter-rater)
  * Validity (concurrent validity against established tools and construct validity)
  Interventions: Other: Traditional physical therapy

INTERVENTIONS:
Other: Traditional physical therapy — Application of laser three times per week in addition to applying deep friction massage, stretching exercises along with the uses of pressure garment.

SUMMARY:
This study uses a mixed-method design combining a quasi-experimental, single-group pre-post intervention with a methodological validation approach.

DETAILED DESCRIPTION:
1. Quasi-experimental, single-group pre-post intervention:

   Participants will receive a standardized physical therapy protocol targeting scar contracture. After intervention, scar extensibility will be measured using traditional tools (Vancouver Scar Scale, tonometer) and a newly developed image-based method.
2. Methodological validation approach: The image-based method will be tested for:

   * Reliability (test-retest, inter-rater)
   * Validity (concurrent validity against established tools and construct validity)

ELIGIBILITY:
Inclusion Criteria:

* History of clinically diagnosed scar contracture following thermal burns.
* Presence of scars (≥6 months post-burn) to ensure stability for accurate assessment.
* Scars located on functionally mobile areas (e.g., limbs) where extensibility impacts daily activities.
* Willingness to undergo a standardized physical therapy intervention.
* Ability to provide informed consent and comply with all study procedures.

Exclusion Criteria:

* Active infection, unhealed wounds, or unstable scars at the assessment site.
* Diagnosed systemic diseases affecting collagen synthesis or wound healing (e.g., scleroderma, uncontrolled diabetes).
* History of experimental or non-standard scar treatment within the last 3 months.
* Severe cognitive impairments or communication barriers that interfere with understanding or participation.
* Pregnant or lactating women, due to hormonal influences on tissue healing and collagen metabolism.
* Concurrent participation in other physical therapy or rehabilitation studies targeting scar management.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-05-04 (Estimated); Study Completion 2025-05-12 (Estimated)

PRIMARY OUTCOMES:
Vancouver Scar Scale (VSS) | Baseline and three months after the intervention
  to evaluate vascularity, pigmentation, pliability, and scar height.
Firmness and pliability at the scar site | Baseline and three months after the intervention
  Tonometry will be used to assess tissue firmness and pliability at the scar site.
Proposed Image-Based Method | Baseline and three months after the intervention
  the scar images before and after the intervention will go through three steps:
  * Image Acquisition: High-resolution digital images of scars will be captured using a standardized protocol (fixed camera settings, lighting, distance).
  * Image Preprocessing: Images will be converted to grayscale, and regions of interest (ROI) manually or automatically defined.
  * Image Analysis: The standard deviation (STD) of pixel intensities within the ROI will be calculated as an indicator of tissue extensibility and collagen fiber cross-linking patterns will be detected and quantified using advanced image processing algorithms.

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa MA Elsayeh, PhD, Principal Investigator — Cairo University
Locations (1):
- Shaimaa Mohamed Ahmed Elsayeh, Cairo, New Cairo, Egypt